CLINICAL TRIAL: NCT02887833
Title: An Exploratory Study to Develop and Evaluate a Simple Bedside Tool for Community Use to Identify Who is Most Likely to Benefit From Palliative Radiotherapy for Cancer Induced Bone Pain: Thermal Testing in Bone Pain (TiBoP)
Brief Title: Thermal Testing in Bone Pain (TiBoP)
Acronym: TiBoP
Status: Completed | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: 16/SC/0260
Record Dates: First submitted 2016-08-29; First posted 2016-09-02 (Estimated); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Cancer Induced Bone Pain; Secondary Malignant Neoplasm of Bone; Toxicity Due to Radiotherapy; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood; Urine
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- XRT for Cancer induced bone pain: Will have community based assessment before and after radiotherapy to assess feasibility of using a clinical biomarker (thermal sensory testing) to predict treatment response
  Interventions: Other: Clinical biomarker (thermal sensory testing)

INTERVENTIONS:
Other: Clinical biomarker (thermal sensory testing) — Thermal sensitivity testing: The area of CIBP and a corresponding unaffected (control) area will be assessed using warm and cool thermal rollers (Rolltemp, Somedic, Sweden). The control area will either be the contralateral side, or an area proximal to the affected site.

SUMMARY:
If cancer spreads to bones it can be very painful, especially when trying to move around. One of the best treatments is radiotherapy, which has to be given in a cancer centre. Even with this treatment, only about half of people will get good pain relief, and that can take up to 6 weeks to work fully. If we know who is unlikely to benefit , then we can explore other forms of pain relief sooner, without having to go through radiotherapy unnecessarily.

We have found that there may be a very simple way to identify patients likely to get good pain relief, using a test of changes in temperature sensation over the painful bone. This study will explore whether this simple bedside test can be used in a community setting to identify which patients suffering from cancer induced bone pain will get good pain relief from radiotherapy.

DETAILED DESCRIPTION:
Bone is the third most common site of metastatic disease, after liver and lung, with ~75 per cent of these patients suffering from related pain. Cancer-induced bone pain (CIBP) remains one of the major clinical challenges in palliative care, with a number of possible reasons for this. Bone pain can have a significant impact on physical, psychological and social functioning (and so overall quality of life). The mechanisms of CIBP are complex and may have unique characteristics that are different from neuropathic and inflammatory pain - this has clear implications for managing CIBP effectively. Current gold standard treatment for CIBP is palliative radiotherapy (XRT). Radiotherapy is the current standard treatment for CIBP, although only 55% of patients will achieve adequate analgesia from palliative radiotherapy, and this can take up to 6 weeks to work. There has been considerable interest in how clinical signs and symptoms in pain translate into underlying mechanisms, and how this may be used to direct treatment more effectively. The clinical assessment of somatosensory processing used for neuropathic pain can be extensive, and burdensome for frail patients.

The investigators have developed a modified assessment for use in patients with cancer, that can be used in a hospital setting. The investigators clinical pilot work used detailed phenotyping of CIBP, to try and better understand underlying mechanisms and detect changes in somatosensory processing. The investigators found that changes in temperature sensitivity may predict pain relief from XRT. Following on from this the investigators propose to develop a simple bedside tool, suitable for use in the community, which will potentially identify patients most likely to benefit from radiotherapy.

Development of this tool requires adequate validation and evaluation so that it can be used as an aid to deciding which patients are more likely to benefit from radiotherapy. In those patients unlikely to benefit, early identification would allow use of other symptom control strategies in the community, minimising the burden of unnecessary hospital attendance, and avoiding the acute pain flare that can occur with XRT.

The investigators hypothesis is that alterations in thermal sensitivity will reflect important changes in underlying pain neurobiology that will make that patient more, or less, likely to get effective analgesia from XRT. Assessment of CIBP There have been recommendations suggested for the use of pain measurement tools and methods in clinical practice to try and include the wider aspects of the pain experience (www.immpact.org). In patients with cancer, it is important to minimise any burden from assessment. We have therefore use a very a simple approach to try and capture the important elements of CIBP and its impact. This consists of a number of validated self report questionnaires (see below), plus a measurement of skin sensitivity to warm and cool (40°C, 25°C), as identified from our previous work as potential predictors of treatment response to XRT.

Self report measures include: the Brief Pain Inventory (BPI); The Short-Form McGill Pain Questionnaire (SF-MPQ-2); the Hospital Anxiety & Depression Scale (HADS); the Distress Thermometer; the EORTC health-related quality of life questionnaire for bone metastases.

Patients with CIBP will be assessed prior to XRT, then at 2, 6 and 12 weeks after XRT.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of cancer with pain related to bony disease (pain ≥4/10 on a numerical pain rating scale);
* due to receive XRT for CIBP;
* outpatient;
* age 18-100;
* able to complete assessment and give written informed consent.

Exclusion Criteria:

* • they are confused or suffering from significant psychiatric illness

  * their condition is unstable or rapidly deteriorating
  * they have any other medical condition that would confound the objectives of the study
  * they who would be adversely affected by study participation. This would include those who are unaware of the presence of progressive disease or who would, in the opinion of the medical team, find completion of the study too burdensome
  * they would be unable to complete the study protocol for any other reason

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer induced bone pain scheduled to undergo palliative radiotherapy for this
Sampling Method: Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of the thermal sensitivity score in CIBP with respect to experiencing a "positive outcome" after XRT | 6 weeks
  A positive outcome is defined as: at least 30% reduction in BPI pain at 6 weeks AND no increase in opioid medication use within 6 weeks AND no toxicity from XRT at 2 weeks.

SECONDARY OUTCOMES:
Sensitivity and specificity of thermal testing with respect to experiencing a positive outcome | 12 weeks
  A positive outcome is defined as: at least 30% reduction in BPI pain at 6 weeks AND no increase in opioid medication use within 6 weeks AND no toxicity from XRT at 2 weeks.
Change in validated self report measures of the pain experience | 2,6,12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Colvin, PhDFRCA FRCP, Principal Investigator — NHS Lothian/ University of Edinburgh; Marie Fallon, MD FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Edinburgh Cancer Centre, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laird BJ, Walley J, Murray GD, Clausen E, Colvin LA, Fallon MT. Characterization of cancer-induced bone pain: an exploratory study. Support Care Cancer. 2011 Sep;19(9):1393-401. doi: 10.1007/s00520-010-0961-3. Epub 2010 Aug 1. PMID 20680354
- [Background] Delaney A, Fleetwood-Walker SM, Colvin LA, Fallon M. Translational medicine: cancer pain mechanisms and management. Br J Anaesth. 2008 Jul;101(1):87-94. doi: 10.1093/bja/aen100. Epub 2008 May 19. PMID 18492671
- [Result] Parker RA, Sande TA, Laird B, Hoskin P, Fallon M, Colvin L. Bayesian methods in palliative care research: cancer-induced bone pain. BMJ Support Palliat Care. 2022 May;12(e1):e5-e9. doi: 10.1136/bmjspcare-2019-002160. Epub 2020 Mar 5. PMID 32139358